CLINICAL TRIAL: NCT03974542
Title: Telephone Outreach by Navigators to Improve Repeat Fecal Occult Blood Testing in Population Colorectal Cancer Screening Programme- a Randomised Control Trial
Brief Title: Telephone Outreach by Navigators to Improve Repeat Fecal Occult Blood Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre for Health Protection, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Grace Wong, Medical Officer, Centre for Health Protection, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CRC
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone outreach (Experimental)
  Interventions: Behavioral: telephone outreach
- control (No Intervention)

INTERVENTIONS:
Behavioral: telephone outreach — The navigator should make at least five (5) attempts to reach the participants on different days (at least one (1) attempt in weekend) and different time slots (at least one (1) attempt each in am, pm and evening). If the navigator only reached voice mail after the 1-month intervention period, a standard script will be read and a contact number will be provided.
  Arms: telephone outreach

SUMMARY:
To conduct a randomised control trial to test the effectiveness of telephone outreach programme to improve the uptake rate of repeat fecal occult blood test in colorectal cancer screening programme.

DETAILED DESCRIPTION:
The colorectal cancer screening programme(CRCSP) adopts a two-tier approach, offering faecal occult blood test (FOBT) by FIT as first line screening followed by colonoscopy examination for cases with positive FIT result. Under the CRCSP, participants with negative or uninformative FIT result in the first round should be re-screened after 24 months.

The objective is to conduct a randomised control trial to test the effectiveness of telephone outreach programme to improve the uptake rate of repeat fecal occult blood test in CRCSP.

ELIGIBILITY:
Inclusion Criteria:

* Participants of CRCSP born between 1949 and 1951 with negative or uninformative FIT result in the first screening round who are due for second rescreening round for at least 4 months but did not turn up for rescreening

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
rescreening of CRC | 2 months
  completion of repeated fecal occult blood test in CRCSP
rescreening of CRC | 5 months
  completion of repeated fecal occult blood test in CRCSP

IPD SHARING:
Plan to Share IPD: No